CLINICAL TRIAL: NCT07316270
Title: SAfety and eFfectiveness of cathetER Ablation for Atrial Fibrillation With Intracerebral Hemorrhage (SAFER-AF)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of Cardiology Department, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS2025246
Record Dates: First submitted 2025-12-15; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: AF - Atrial Fibrillation; ICH - Intracerebral Hemorrhage
MeSH Terms: conditions — Atrial Fibrillation; Cerebral Hemorrhage | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care Group (Active Comparator)
  Interventions: Drug: Usual Care
- Catheter Ablation Group (Experimental)
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — All patients undergo pulsed field ablation, followed by low-dose rivaroxaban for 1 month. For patients with paroxysmal atrial fibrillation (AF), an ablation strategy based on bilateral pulmonary vein isolation (PVI) is adopted. For patients with persistent AF, PVI plus ethanol infusion of the vein of Marshall and linear ablation (mitral isthmus, cavotricuspid isthmus, and left atrial roof) strategy is recommended. Other additional ablation strategies are determined by the operator. Anticoagulation therapy is discontinued after 1 month if no AF is detected during patient monitoring.
  Arms: Catheter Ablation Group
Drug: Usual Care — The use of antithrombotic therapy is at the discretion of the treating physician.
  Arms: Usual care Group

SUMMARY:
SAFER-AF is an investigator-initiated, multicenter, open-label, parallel-group trial comparing catheter ablation versus usual care in patients with atrial fibrillation and intracerebral hemorrhage.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) increases the risk of stroke, heart failure, and mortality. Oral anticoagulation is the standard treatment for preventing thromboembolism, but it also raises the risk of bleeding. About 20-25% of patients with intracerebral hemorrhage (ICH) have AF. Previous randomized trials indicate that restarting anticoagulation may prevent ischemic stroke, but increase risk of recurrent ICH. Catheter ablation is the first-line rhythm control strategy that reduce thromboembolic risk by maintaining sinus rhythm and potentially reducing the need for long-term anticoagulation. Pulsed field ablation (PFA) uses electroporation to ablate the myocardium by electroporation with high tissue specificity and may shorten the required anticoagulation period.

The SAFER-AF trial is a prospective, multicenter, open-label randomized controlled trial enrolling 646 AF patients with previous spontaneous ICH, investigating whether catheter ablation provides superior long-term net clinical benefit compared with usual care. Participants will be randomized 1:1 to catheter ablation versus usual care, with a minimum follow-up of 2 years. Patients in catheter ablation group will undergo PFA, followed by low-dose direct oral anticoagulants for 1 month. The primary endpoint is the composite of all-cause mortality, all-cause stroke (ischemic or hemorrhagic), and systemic embolism. SAFER-AF aims to define a safer, individualized therapeutic pathway balancing ischemic protection and hemorrhagic risk, ultimately improving survival and long-term outcomes for AF patients with ICH.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Between 14 Days and 12 Months After Spontaneous Intracerebral Hemorrhage
3. Able to Access Intracerebral Hemorrhage Imaging Data
4. ECG indicating the presence of atrial fibrillation
5. CHA₂DS₂-VA Score ≥ 2
6. Willing to undergo randomization and able to complete follow-up as required

Exclusion Criteria:

1. Atrial fibrillation secondary to clearly reversible causes (e.g., hyperthyroidism, hypokalemia, etc.)
2. Fully dependent (modified Rankin Scale [mRS] score > 4)
3. Uncontrolled hypertension (systolic blood pressure > 160 mmHg)
4. Presence of uncontrolled active bleeding
5. Presence of active infection requiring antibiotic treatment
6. End-stage renal failure or receiving dialysis treatment
7. Presence of liver failure
8. Untreated coronary artery disease with indication for revascularization
9. Presence of intracardiac masses, thrombi, etc., as evaluated by transthoracic echocardiography or transesophageal echocardiography
10. Expected life expectancy < 1 year (e.g., advanced malignant tumors, etc.)
11. Pregnant, lactating, or women planning to become pregnant
12. Presence of psychological or psychiatric disorders that prevent understanding or cooperation with the study
13. Other conditions deemed unsuitable for participation in the study by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Composite of All-Cause Mortality, All-Cause Stroke, and Systemic Embolism | 48 months

SECONDARY OUTCOMES:
Stroke and Systemic Embolism | 48 months
Cardiovascular death | 48 months
Ischemic Stroke | 48 months
Intracerebral Hemorrhage | 48 months
ISTH Major Bleeding | 48 months
Change in quality of life assessed by the Atrial Fibrillation Effect on QualiTy of life (AFEQT) questionnaire | 48 months
  The Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire is a disease-specific, patient-reported outcome measure assessing health-related quality of life in patients with atrial fibrillation. The overall AFEQT score ranges from 0 to 100, with higher scores indicating better quality of life.
Change in health-related quality of life assessed by the EQ-5D-5L questionnaire | 48 months
  The EQ-5D-5L (EuroQol five-dimension, five-level) questionnaire is a standardized, generic measure of health-related quality of life. It consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity. Health states are converted into a single index value using a country-specific value set, with higher index values indicating better health-related quality of life.
Change in cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | 48 months
  The Montreal Cognitive Assessment is a 30-point cognitive screening tool assessing multiple cognitive domains. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Change in cognitive function assessed by the Mini-Mental State Examination (MMSE) | 48 months
  The Mini-Mental State Examination is a 30-point questionnaire used to assess global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xiamen Cadiovascular Hospital, Xiamen, Fujian
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No